CLINICAL TRIAL: NCT07330414
Title: CUHK Achilles Tendon Disorder Registry
Acronym: AT Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor of Orthopaedics and Traumatology, CUHK Head of the Foot and Ankle Team / Honorary Associate Consultant, Prince of Wales Hospital Specialist in Orthopaedics and Traumatology, CUHK Medical Centre, Chinese University of Hong Kong
Other Study IDs: 2025.699
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Achilles Tendon Injury; Achilles Tendon; Achilles Tendon Pain
Keywords: Achilles tendinopathy; Achilles tendon rupture; Achilles tendinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Healthy individuals without any Achilles tendon injury
- Achilles tendon disorder group: Individuals with any Achilles tendon disorder

SUMMARY:
This is a long-term research registry for patients with Achilles tendon disorders (like tears, chronic pain, or ruptures) as well as healthy adults without tendon problems. The goal is to collect detailed information over time to understand which treatments work best for different people, identify risk factors for injury, and improve overall care. Adults over 18, both with and without Achilles tendon conditions, are eligible to join. Participants will attend several assessment visits at the Prince of Wales Hospital over the first year (at the start, 6 weeks, 3, 4, 6, and 12 months) for physical tests, ultrasounds, and questionnaires. After the first year, follow-up continues with annual online questionnaires for up to five years. The main measure is a standard questionnaire about tendon pain and function (VISA-A). The study aims to use this information to guide better, more personalized rehabilitation strategies, improve patient outcomes, and reduce long-term disability. All participation is voluntary and requires written consent.

DETAILED DESCRIPTION:
This is a prospective, longitudinal Achilles Tendon Registry study. The registry is conceived as a foundational cohort study designed to systematically address critical evidence gaps in the management of Achilles tendon pathologies. The Achilles tendon, while robust, is susceptible to a spectrum of disorders including acute ruptures and chronic tendinopathies, often summarized colloquially as the "Achilles heel." Current clinical management strategies for these conditions are characterized by heterogeneity, largely due to a paucity of high-quality, longitudinal comparative effectiveness data. This registry aims to mitigate this gap by creating a centralized repository of standardized, prospective data, thereby enabling rigorous evaluation of treatment outcomes, prognostic factors, and long-term sequelae.

The primary objective is to establish a comprehensive, prospectively enrolled cohort of individuals with Achilles tendon disorders, complemented by a cohort of asymptomatic controls, to facilitate comparative and predictive analyses. The study is explicitly designed to answer three pivotal research questions. First, it will investigate the prognostic influence of baseline structural and vascular status of the tendon, as quantified by ultrasonographic and elastographic metrics, on functional recovery. Second, it will assess whether a pre-existing diagnosis of Achilles tendinopathy constitutes a significant risk factor for subsequent acute tendon rupture. Third, it will analyze differential treatment responsiveness, aiming to identify which patient subgroups, defined by specific baseline characteristics, demonstrate optimal outcomes with specific treatment modalities.

The study methodology is that of a prospective, single-center cohort study to be conducted at the Prince of Wales Hospital in Hong Kong. The target sample size is a minimum of 500 participants, to be consecutively enrolled from 2025 to 2028. The participant pool will include adults over the age of 18 with a diagnosis of an Achilles tendon disorder, as well as asymptomatic control participants without tendon pathology. Key exclusion criteria encompass any comorbid physical or psychological condition that would impair the ability to complete study assessments or provide informed consent, and concomitant diseases that severely affect lower limb function (e.g., severe osteoarthritis, prior amputation, active inflammatory arthritis, or paralysis).

The follow-up protocol is structured into intensive initial and long-term phases. All participants will undergo comprehensive in-person assessments at baseline, 6 weeks, 3 months, 6 months, and 1 year post-enrollment. These assessments constitute the core data collection points and encompass a multi-modal battery of outcome measures. Following the initial 1-year follow-up, the protocol transitions to long-term monitoring, wherein all self-reported outcome measures will be collected annually via online questionnaires at years 2, 3, 4, and 5.

The primary outcome measure is the Victorian Institute of Sports Assessment-Achilles (VISA-A) questionnaire, a validated, disease-specific patient-reported outcome tool scored from 0 to 100. A comprehensive suite of secondary outcome measures will be collected to provide a holistic assessment. These include patient-reported outcomes such as the Numeric Pain Rating Scale (NPRS) and the Foot and Ankle Outcome Score (FAOS). Functional and physical performance measures are integral and consist of the Achilles Tendon Resting Angle (ATRA), calf muscle strength quantified via hand-held dynamometry, the heel raise endurance test, and a one-legged counter-movement jump test performed on a pressure mat. Biomechanical analysis includes foot pressure distribution assessment and treadmill-based gait analysis using a Zebris system.

A central and rigorous component of the assessment protocol is ultrasonographic evaluation, performed at all in-person time points using a standardized imaging protocol. Key sonographic parameters include tendon thickness and cross-sectional area, neovascularity scored via the Öhberg scale, and tendon elasticity quantified by shear wave elastography (SWE) to measure stiffness in kilopascals. Supplementary advanced imaging modalities may be employed in subsets of participants, including photoacoustic ultrasound (PAUS) for quantifying tendon oxygenation and vascularity, and infrared thermography for measuring superficial tendon temperature.

Data management and security are paramount. All collected data, including personally identifiable information and consent forms, will be stored under strict physical and electronic security protocols. Physical documents will be kept in locked cabinets, and electronic data on password-protected computers. Data entry will employ a double-entry method with range checks to ensure accuracy. The final analysis dataset will be de-identified. Access to identifiable data is restricted to authorized trial team members. De-identified data may be shared with external researchers upon reasonable request, execution of a data sharing agreement, and following approval by the relevant ethics committee.

Statistical analysis will be performed using SPSS software (version 28.0) with a two-sided alpha level of 0.05. Analytical strategies are tailored to the research questions. Multivariable linear or logistic regression will evaluate associations between baseline metrics and outcomes (Q1). Cox proportional hazards or logistic regression models will assess the risk of rupture associated with pre-existing tendinopathy (Q2). To identify differential treatment effects (Q3), regression models will incorporate interaction terms between patient subgroups and treatment types, with subsequent stratified analysis if interactions are significant. Missing data will be handled using multiple imputation techniques, and sensitivity analyses will be conducted. An interim analysis for safety monitoring will be performed after 20% of participants complete the 1-year follow-up.

The study will be overseen by a Trial Steering Committee comprising the Principal Investigator, orthopaedic surgeons, research assistants, and a biostatistician from the research team. The committee is responsible for monitoring study progress, participant recruitment, and data collection. An independent annual audit of trial conduct will be performed by an auditor from the Joint Chinese University of Hong Kong - New Territories East Cluster Clinical Research Ethics Committee. All protocol amendments will require prior ethics committee approval and will be communicated to participants and registered publicly.

The study is conducted under the auspices of the Department of Orthopaedics and Traumatology, Faculty of Medicine, The Chinese University of Hong Kong. No external funding sources or sponsors have been declared at this protocol stage. All investigators have declared no competing interests. Participants will not receive financial incentives. Provisions for harm are established: any participant experiencing an adverse effect directly attributable to the study procedures will receive appropriate medical care at the Prince of Wales Hospital at no additional cost, with compensation handled per institutional and ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)

Exclusion Criteria:

* Any physical or psychological comorbidity that would impair the ability to complete study assessments (e.g., significant neurological deficits) or preclude the provision of informed consent.
* Concomitant diseases that severely affect lower limb function or assessment (e.g., severe osteoarthritis of the knee or hip, prior lower limb amputation, peripheral vascular disease, active rheumatoid arthritis, lower limb paralysis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hong Kong Residents
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment (VISA-A) | From enrollment to 5 years after baseline assessment
  The primary outcome measure will be the Victorian Institute of Sport Assessment (VISA-A) questionnaire, available in either the original English or validated Chinese version, depending on the participant's native language. This specific scoring system developed for the Achilles tendon is the most widely used score for clinical Achilles research. The VISA-A is scored on a scale of 0 to 100; lower scores indicate more severity of symptoms, while a score of 100 indicates a healthy and pain-free Achilles tendon.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | From enrollment to 5 years after baseline assessment
  The Numeric Pain Rating Scale (NPRS; 0-10, where 10 represents maximum pain) will be used to assess pain levels, as pain is the primary symptom of midportion Achilles tendinopathy. Participants will report their "Worst pain during sports in the past two weeks," "Worst pain during daily activities in the past two weeks."
Foot and Ankle Outcome Scores (FAOS) | From enrollment to 5 years after baseline assessment
  The FAOS is a validated patient-reported scoring system used for general foot and ankle problems. It is split into five categories: symptoms, pain, daily activities, sporting function, and quality of life. Scores range from 0 to 100, with 0 being the lowest and 100 being the highest.
Achilles tendon resting angle (ATRA) | From enrollment to 1 year after baseline assessment
  The ATRA will measure participants' tendon length/tension. Participants should be positioned in a prone position with the knee flexed to 90 degrees. The assessor will use a dynamic joint goniometer to measure the angle at which the foot passively falls.
Royal London hospital test | From enrollment to 1 year after baseline assessment
  The Royal London Hospital Test is used to help diagnose mid-portion Achilles tendinopathy. The patient lies prone with the foot relaxed, and the examiner palpates the most tender spot on the Achilles tendon. The patient then moves the ankle through dorsiflexion and plantarflexion. A positive test occurs if tenderness decreases during dorsiflexion.
Calf Muscle Strength | From enrollment to 1 year after baseline assessment
  The hand-held dynamometer will be used to quantify isometric muscle strength during ankle dorsiflexion and plantarflexion. Participants will maintain maximal isometric contraction for 3 seconds. Three trials will be recorded for each movement, with 30-second rest intervals between trials to prevent fatigue.
Heel raise test | From enrollment to 1 year after baseline assessment
  Participants will be instructed to keep the knee straight and rise as high as possible on the toes each time until fatigue. Participants can place two fingertips per hand on the wall to maintain balance. The rhythm will be set at a frequency of 30 heel rises per minute by following a metronome. Total test duration (in seconds) will be recorded
Jump test | From enrollment to 1 year after baseline assessment
  Participants will perform three one-legged counter-movement jumps on a pressure mat (Tekscan, USA) with jump height (cm) calculated from flight time. After demonstration and submaximal practice jumps, the patient executed maximal jumps from a standing position by rapidly squatting (flexing knee/hip/ankle) before exploding upward. The highest jump was recorded, with NPRS-reported Achilles tendon pain immediately post-test.
Foot pressure distribution | From enrollment to 1 year after baseline assessment
  In foot pressure distribution examination, the scan (Tekscan, USA) will be masked and divided the foot into eight regions including both forefoot, midfoot and hindfoot: hallux, lesser toes, lateral and medial forefoot, lateral and medial midfoot, lateral and medial hindfoot. Peak pressure and impulse in each region will be calculated to see the before-and-after change. Additionally, the centre of pressure excursion index (CPEI) will also be calculated to which reflects the excursion of the centre of pressure. The first and last points of a centre of pressure curve will be connected to construct a line measured in the distal tertile of the foot and normalized by the foot's width.
Zebris Treadmill Gait and Stance Analysis | From enrollment to 1 year after baseline assessment
  The Zebris is a treadmill equipped with advanced pressure sensors designed to analyze gait and stance. Subjects were instructed to walk barefoot on the treadmill at their comfortable pace while maintaining a natural walking pattern. During the test, the pressure distribution across the plantar surface of the feet was recorded, capturing dynamic data such as force, timing, and spatial parameters of each step, which ensures precise measurement of walking and stance characteristics, providing valuable insights into balance, weight distribution, and movement symmetry for clinical or research purposes.
Tendon oxygenation and vascularity | From enrollment to 1 year after baseline assessment
  The pathological tendon's oxygenation and vascularity were quantified using a multiwavelength photoacoustic ultrasound (PAUS) system equipped with a 7Hz probe and dual-wavelength LED sources (850nm/750nm). The participant assumes a prone position with heels extended beyond the examination table. The probe is positioned on the target tendon, with mode-specific presets selected ("Deep PA" for vascularity at 850nm; "Deep Oxy" for oxygenation at 750nm). Each 20-second acquisition captures 200 frames, with two repeated scans per mode to ensure data reliability.
Achilles Ultrasonography- Tendon Thickness | From enrollment to 1 year after baseline assessment
  Using B-mode ultrasound scanning, the probe is moved from the medial to the lateral aspect of the Achilles tendon until a planar image of the Achilles tendon is clearly shown. The probe was adjusted straight perpendicular to the tendon fibres. A greyscale sonogram is acquired, and the tendon thickness is measured at the maximum thickness point and at 2, 4, 6 cm proximal to the insertion. Less than 5.3 mm was considered a healthy value for the Achilles tendon.
Achilles Ultrasonography - Tendon vascularity | From enrollment to 1 year after baseline assessment
  Vascularity will be documented using the Ohberg score. Using the Doppler mode on the ultrasound machine, the transducer is placed vertically to obtain a sagittal view of the softest area of the Achilles tendon. Pressure on the skin from the transducer should be kept to a minimum to prevent occlusion of blood vessels. The colour box is focused on the dorsal aspect of the tendon. The assessor will spend one minute exploring the blood flow over the tendon to find the area of maximum Doppler flow. After locating the area, sonograms are taken to determine the Öhberg score. The Öhberg score ranges from 0 to 3 points. In this scoring system, the score is defined as 0 (no neovascularisation, healthy), 1 (mild neovascularisation with a few single vessels), 2 (moderate neovascularisation with a moderate number of mostly transverse vessels), and 3 (multiple, mostly transverse vessels distributed throughout the depth of the tendon). Higher scores indicate more Doppler blood flow in the periten
Achilles Ultrasonography - Tendon elasticity | From enrollment to 1 year after baseline assessment
  Shear wave elastography (SWE) can be used to quantify soft tissue stiffness. Once the optimal scan plane of the tendon is determined, the SWE function is activated. It enters penetration mode and the measured stiffness range is normalized to 0-600 kPa. The SWE color card (H × W: 1.4 cm × 1.3 cm) is placed immediately above the upper edge of the calcaneus. After the color signal stabilized for five seconds, the elastogram was recorded and stored. Tendon stiffness was measured using a Q-box stiffness meter. Depending on the size of the tendon, the diameter of the circular measuring area (Q-box) is set to 2 mm, which covers the Achilles tendon and excludes other adjacent soft tissues. The Q-box is located in the center of the maximum thickness point and 2, 4, 6 cm proximal to the calcaneal insertion site. For each Q-box, the average tendon stiffness (in kPa) is measured.
Thermographic tendon temperature | From enrollment to 1 year after baseline assessment
  Participants will be advised to avoid physical exercise and hot baths before the procedure to ensure data reliability. Each participant will rest in a seated position for 10 minutes followed by 2 minutes without socks. The room will be maintained at 20-24°C. The infrared camera will be positioned one meter from the participant, using a ThermaCam FLIR-T8210. Images will be analyzed with ThermaCAM Researcher Pro 2.8 SR-1 software, and a rectangular area covering the Achilles tendon will be used for temperature assessment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ko VM, He X, Fu SC, Yung PS, Ling SK. Clinical effectiveness of pulsed electromagnetic field therapy as an adjunct treatment to eccentric exercise for Achilles tendinopathy: a randomised controlled trial. Trials. 2023 Jun 12;24(1):394. doi: 10.1186/s13063-023-07434-6. PMID 37308969
- [Background] Ko VM, Chen SC, He X, Fu SC, Franco-Obregon A, Yung PS, Ling SK. Short-term Effects of Pulsed Electromagnetic Field Therapy for Achilles Tendinopathy: A Randomized Controlled Trial. Orthop J Sports Med. 2024 Nov 12;12(11):23259671241284772. doi: 10.1177/23259671241284772. eCollection 2024 Nov. PMID 39534390

DOCUMENTS (1):
  • Study Protocol (2025-10-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT07330414/Prot_000.pdf